CLINICAL TRIAL: NCT06604130
Title: Plasma Exosome RNA Combination for Diagnosing Prostate Cancer: a Prospective, Multicenter Diagnostic Trial
Brief Title: Plasma Exosome RNA to Diagnose Prostate Cancer
Acronym: exo-PRECISE
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Xijing Hospital (Other)
Collaborators: Shaanxi Provincial People's Hospital (Other); Yan'an University Affiliated Hospital (Other); Weinan Central Hospital (Other); The Second Affiliated Hospital of Shaanxi University of Chinese Medicine (Unknown); Affiliated Hospital of Qinghai University (Other); General Hospital of Ningxia Medical University (Other); LanZhou University (Other); Air Force 986 Hospital (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Diagnostic
Other Study IDs: KY20242271-C-1; NSFC(China) (Other Grant/Funding Number: National Natural Science Foundation of China)
Record Dates: First submitted 2024-09-13; First posted 2024-09-19 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Prostate Cancer
Keywords: Prostate cancer; RNA; Diagnosis; Combination
MeSH Terms: conditions — Prostatic Neoplasms; Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- The experimental arm receiving diagnosis from serum RNA combination (Experimental)
  Interventions: Diagnostic Test: Prostate cancer screening decision

INTERVENTIONS:
Diagnostic Test: Prostate cancer screening decision — The subjects would receive serum PSA test.

SUMMARY:
The aim of the present study is to investigate a RNA combination to diagnose prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Blood prostate-specific antigen PSA>4ng/dl;
2. Patients suspected of having prostate cancer through clinical symptoms, digital rectal examination, ultrasound examination, magnetic resonance imaging, and PSMA PET/CT examination.
3. The patient is willing to undergo prostate biopsy.

Exclusion Criteria:

1. Previous diagnosis of prostate cancer through prostate biopsy;
2. History of other malignant tumors in the past two years;
3. According to the research physician's judgment, serious complications may occur and affect the normal conduct of the experiment

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1600 (Estimated)
Dates: Start 2021-03-12 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
The diagnostic efficacy of plasma exo-RNA panel alone in diagnosing PCa | The time of prostate biopsy and after 6 months follow-up
  The primary outcome is to investigate a plasma-exosome RNA panel in diagnosing prostate cancer and evaluate its sensitivity and specificity in diagnosing PCa.
  Descriptive statistics were calculated and presented as the frequency (percentage) for categorical variables, the mean (standard deviation) for continuous variables with a normal distribution, and the median (quartile) for continuous variables with a skewed distribution. Two-sample t-tests were used to assess continuous variables with a normal distribution, and the Wilcoxon signed-rank test was used to assess continuous variables with a skewed distribution. The Mann-Whitney U test was used to compare means from two samples. The correlation between two samples was analyzed by Spearman's ρ test. The receiver operating characteristic (ROC) curve was used to determine the cutoff value of exo-RNA panel for diagnosing patients with PCa.

SECONDARY OUTCOMES:
Diagnostic efficacy of plasma exo-RNA panel in diagnosing csPCa, insignPCa and its comparison with other imaging methods or blood tests | The time of prostate biopsy and after 6 months follow-up
  The secondary outcome is to evaluate the positive predictive value (PPV), negative predictive value (NPV) and accuracy of exo-RNA panel in detection of PCa; to evaluate the perforamce of exo-RNA panel in identifying grade group 2 (GG2) or higher clinically significant prostate cancer (csPCa) tumors and compare the diagnostic performance of the plasma-exosome RNA panel with other imaging methods or blood tests in identifying prostate cancer patients; Whether the exo-RNA panel could predict the PCa patients with higher Gleason score (GS).
  The comparison between diagnostic performance of exo-RNA panel and other imaging or blood tests is performed in ROC curves. The ICC analysis was performed by reliability analysis. All statistical analyses were conducted using IBM SPSS statistics software, version 23.0 (IBM, Inc., Chicago, IL, USA) and GraphPad Prism software, version 8.0 (GraphPad Software, Inc., La Jolla, CA, USA).

CONTACTS AND LOCATIONS:
Locations (9):
- China (9):
  - The First Hospital of Lanzhou University, Lanzhou, Gansu
  - General Hospital of Ningxia Medical University, Yinchuan, Ningxia
  - Qinghai University Affiliated Hospital, Xining, Qinghai
  - Weinan Central Hospital, Weinan, Shaanxi
  - Shaanxi Provincial People's Hospital, Xi'an, Shaanxi
  - Xijing 986 Hospital, Xi'an, Shaanxi
  - Xijing Hospital, Xi'an, Shaanxi
  - The Second Affiliated Hospital of Shaanxi University of Chinese Medicine, Xianyang, Shaanxi
  - Affiliated Hospital of Yan'an University,, Yan’an, Shaanxi

IPD SHARING:
Plan to Share IPD: Undecided
The subjects may not disclose their IPD totally or partly.